CLINICAL TRIAL: NCT06180473
Title: Evaluation of Tolerability, Efficacy and Adherence to Treatment With Wynzora Cream in Patients With Psoriasis Previously Treated With Enstilar Foam.
Brief Title: Evaluation of Tolerability, Efficacy and Adherence to Treatment With Wynzora Cream
Acronym: psowyn
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6131
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2023-12

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — PPQ, TTAQ PTCS

SUMMARY:
The primary objective is to assess with the PPQ questionnaire the patient preference for Wynzora compared with therapy carried out previously with Enstilar spray foam. Secondary objectives Assess satisfaction with the treatment. Assess adherence to therapy. Evaluate the impact of various clinical and demographic factors on treatment adherence. Evaluate the efficacy of Wynzora cream therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age, of either sex;
* Patients diagnosed with mild-to-moderate psoriasis (PASI and BSA <10) requiring monotherapy topical with Wynzora;
* Patients who have stopped treatment with Enstilar foam for any reason for at least 30 days; and
* Patients whose medical records are accessible and record all demographic parameters, anthropometric and clinical parameters during the treatment period
* Signature of written informed consent;

Exclusion Criteria:

* Patients with palmoplantar, inverse, erythrodermic, guttate, and scalp psoriasis.
* Patients who are taking concomitant systemic therapies for psoriasis, such as. cyclosporine, methotrexate, acitretin, phototherapy or biologic therapies.
* Women who are pregnant or planning to become pregnant.
* Patients with disabilities or other motor problems that could complicate self-medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with psoriasis will be enrolled, who will be according to clinical practice will be prescribed treatment with Wynzora cream for 30 consecutive days, referring to the Dermatology and Venereology outpatient clinics of the Fondazione Policlinico Universitario A. Gemelli, IRCCS Rome
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
preference of wynzora cream | 1 month
  Percentage of patients who prefer treatment with Wynzora compared with treatment with Enstilar at week 4 of use; preference for Wynzora will be assessed by considering a score of 3 or higher on question 5 of the PPQ questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Agostino Gemelli, Rome, Italy